CLINICAL TRIAL: NCT00792376
Title: "NSAIDs in Acute Achilles Tendinopathy: Effect on Pain Control, Leg Stiffness and Functional Recovery in Athletes"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Argentine Tennis Association (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Javier Maquirriain, MD, Argentine Tennis Association
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00045-2008; 1-47-12225-05-1
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Achilles Tendinopathy
Keywords: NSAID; tendon; pain; stiffness; Achilles
MeSH Terms: conditions — Pain | interventions — Etoricoxib; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- etoricoxib (Experimental): etoricoxib (ETO) group (n=28) treated with etoricoxib 120 mg/day orally for 7 days
  Interventions: Drug: etoricoxib; Drug: diclofenac
- diclofenac (Active Comparator): diclofenac (DIC) group (n=28) received diclofenac 150 mg/day/7 days orally.
  Interventions: Drug: diclofenac

INTERVENTIONS:
Drug: etoricoxib — etoricoxib (ETO) group (n=28) treated with etoricoxib 120 mg/day orally for 7 days
  Arms: etoricoxib
Drug: diclofenac — diclofenac (DIC) group (n=28) received diclofenac 150 mg/day/7 days orally.

SUMMARY:
The purpose of this study is to evaluate etoricoxib efficacy in pain control, leg stiffness and functional recovery of patients suffering acute Achilles tendinopathy.

It is hypothesized that etoricoxib (120mg orally/day/7 days) efficacy is not inferior to diclofenac (150mg orally /day/7 days) for pain control in subjects suffering acute Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they are male between 18 and 50 years of age and they suffer acute Achilles tendinopathy (<2 weeks). Diagnosis of Achilles tendinopathy is made by means of activity-related achillodynia, morning stiffness or pain, painful one-legged jumping test, tenderness and decreased sports performance (26). Subjects' age, race, affected tendon (right, left), activity, height and weight will be recorded.

Exclusion Criteria:

* Patients are excluded from the study if they have:
* Prior lower limb surgery or major trauma.
* Bilateral Achilles tendinopathy.
* History of lower limb radiculo-neuropathy or miopathy.
* Hypersensitivity to any NSAIDs.
* Used analgesic agents (NSAIDs, salicilates, narcotic) within 1 week
* Concurrent medical/arthritic disease (e.g. gout, lupus, rheumatoid arthritis).
* Other concurrent medical conditions including diabetes, hypertension, angina or congestive heart failure, ischaemic cardiopathy, malabsorption, morbid - Personal history of renal dysfunction, hepatic dysfunction or anemia
* Used corticosteroids, clopidogrel bisulphate, rifampin, quinolon antibiotics, antiepileptics, muscle relaxants, warfarin, ticlopidine, glucosamine, condroitin sulphate for < 6 months prior to the study start. Patients taking low dose aspirin (100 mg) for cardioprotective benefit will be also excluded. Any other medication consumption will be considered by the investigator and the Ethical Committee.
* Any other condition which, in the opinion of the investigator, could confound the study results or pose a risk to the patient (for example, co-morbid conditions for which NSAIDs are contraindicated).
* History of psychotic illness, dementia or depression
* History of drug or alcohol abuse or dependence.
* Participated in any previous NSAIDs study and received active treatment, or in an investigational trial within 30 days prior to the first visit.
* Inability to communicate or to cooperate with the investigator.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The pre-defined primary efficacy endpoint of the study is a 100-mm pain visual analog scale (P-VAS), where 0= no pain; 100= extreme pain. | 1 week

SECONDARY OUTCOMES:
The secondary study endpoints includes: the VISA-A Questionnaire, the Achilles Tendinopathy Scoring System (ATSS), PGART using a 5-point Likert scale and leg functional stiffness. | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Argentine Tennis Association, Buenos Aires, Argentina